CLINICAL TRIAL: NCT02508974
Title: Prevalence and Impact of Hospital Malnutrition on Associated Outcomes
Brief Title: Prevalence of Hospital Malnutrition in Adult Patients
Status: Completed | Type: Observational
Sponsor: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Prof Renee Blaauw, Professor, University of Stellenbosch
Other Study IDs: N14/06/061
Record Dates: First submitted 2015-05-27; First posted 2015-07-27 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Malnutrition of patients on admission to hospitals are estimated to be as high as 60%, although the prevalence varies between countries. The impact of malnutrition on patient recovery and discharge is severe, with extensive cost implications. This study aims to assess the prevalence of at risk for malnutrition among adult patients admitted to hospital across 3 countries on the African continent.

DETAILED DESCRIPTION:
The prevalence of malnutrition on admission to hospital varies between 15-60%. Knowing the extent of the problem and identifying at-risk patients should be a priority task since malnutrition is associated with increased hospital-related complications; longer length of stay, increased costs related to treatment and higher mortality. Post discharge, malnourished patients have also been linked to more frequent re-admissions, higher morbidity and mortality. Various screening tools are available, including the Nutrition Risk Screening-2002 recommended by European Society for Clinical Nutrition and Metabolism as the preferred screening tool for malnutrition in hospitals in Europe. ASPEN recommends a more comprehensive evaluation and diagnosis procedure. In South Africa, and the rest of Africa, nutritional screening is not routinely done and the investigators do not have any reliable national statistics indicating the extent of the problem. The aim of this study is to determine the prevalence of malnutrition on admission to hospital and to identify the impact thereof on relevant outcomes. Two different internationally recognised tools will be used and validated for the African context. In this multi-country, multi-centre descriptive cross-sectional study 3 hospitals in South Africa, 1 in Ghana and 2 in Kenya will be included. Adult patients (n=400 per hospital) will be screened on admission and at discharge and relevant outcomes (in-hospital and 3-month post-discharge) will be charted. A 50% sub-sample will be used to validate the 2 instruments.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years of age
* Males and females
* Admitted to hospital within the past 48 hours
* Conscious
* Informed consent provided

Exclusion Criteria:

* Paediatric patients younger than 18 years
* Pregnant and lactating females
* Patients admitted to ICU, burns or relevant acute care wards
* Patients admitted to psychiatry or eating disorders units
* Patients on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to the hospitals (3 in South Africa [Tygerberg Academic Hospital, Cape Town; Grootte Schuur Academic Hospital, Cape Town; Chris Hani Baragwanath Hospital, Johannesburg]; 2 in Kenya [Aga Khan University Hospital, Nairobi; Mbagathi district hospital, Nairobi] and 1 in Ghana [Korle Bu Teaching Hospital, Accra]) during the defined study periods will be eligible for inclusion in the study.
Sampling Method: Probability Sample
Enrollment: 2126 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in prevalence of risk for malnutrition during the period of hospitalization | Baseline; day 28
  Baseline (Admission) data will be gathered during to the first 48 hours after hospital admission. Discharge data (Day 28) is collected on day of actual discharge or on day 28 of hospitalization if patient is staying in hospital longer than that. A NRS-2002 score greater than 3 indicates risk for malnutrition.

SECONDARY OUTCOMES:
Association between risk for malnutrition and in-hospital and post-discharge nutritional / medical indicators | Baseline; day 28 and Day 90
  Baseline (Admission) data will be gathered during to the first 48 hours after hospital admission. Discharge data (Day 28) is collected on day of actual discharge or on day 28 of hospitalization if patient is staying in hospital longer than that. Post discharge data will be gathered 3 months after hospital discharge i.e. day 90 (again within a 48 hour period). Nutritional indications refer to weight changes (gain or loss) and changes in appetite (improved, no change or decreased). Medical indicators refer to nr of new complications requiring medical treatment, mortality or re-hospital admission.A NRS-2002 score greater than 3 indicates risk for malnutrition.
Number of patients obtaining similar screening scores as a measure of relative validity of the different screening tools used against each other | Baseline and day 28
  Baseline (Admission) data will be gathered during to the first 48 hours after hospital admission. Discharge data (Day 28) is collected on day of actual discharge or on day 28 of hospitalization if patient is staying in hospital longer than that. A good validity will be indicated by a sensitivity and specificity of more than 80%.

CONTACTS AND LOCATIONS:
Overall Officials: Renee Blaauw, PhD, Principal Investigator — University of Stellenbosch
Locations (1):
- Tygerberg Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Undecided